CLINICAL TRIAL: NCT01817699
Title: A Factorial Randomized Controlled Trial of Correcting Anemia and Native Vitamin D Supplementation in Kidney Transplant Recipients
Brief Title: Correcting Anemia and Native Vitamin D Supplementation in Kidney Transplant Recipients
Acronym: CANDLE-KIT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The independent Data Monitoring Committee recommended an early termination.
Sponsor: CANDLE-KIT Trial Study Group (Other)
Collaborators: Chugai Pharmaceutical (Industry); Japanese Society for the Promotion of Science (Other); The Japan Kidney Foundation (Other); Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CKDR-001; UMIN000009970 (Registry Identifier: UMIN Clinical Trials Registry)
Record Dates: First submitted 2013-03-21; First posted 2013-03-25 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Kidney Transplantation; Anemia; Vitamin D Deficiency; Renal Insufficiency, Chronic
Keywords: Cholecalciferol; Methoxy polyethylene glycol-epoetin beta; Hematinics; Bone Diseases, Metabolic; Neoplasms; Cardiovascular Diseases; Graft Rejection
MeSH Terms: conditions — Anemia; Vitamin D Deficiency; Renal Insufficiency, Chronic; Bone Diseases, Metabolic; Neoplasms; Cardiovascular Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low Hb target without cholecalciferol (No Intervention): Target Hemoglobin level: ≥9.5 and <10.5 g/dL
- Low Hb target with cholecalciferol (Active Comparator): Target Hemoglobin level: ≥9.5 and <10.5 g/dL Cholecalciferol: 1,000 IU/day
  Interventions: Dietary Supplement: cholecalciferol
- High Hb target without cholecalciferol (Active Comparator): Target Hemoglobin level: ≥12.5 and <13.5 g/dL
  Interventions: Other: High Hb target
- High Hb target with cholecalciferol (Experimental): Target Hemoglobin level: ≥12.5 and <13.5 g/dL Cholecalciferol: 1,000 IU/day
  Interventions: Other: High Hb target; Dietary Supplement: cholecalciferol

INTERVENTIONS:
Other: High Hb target — 25 to 250 μg of methoxy polyethylene glycol epoetin beta (Mircera®, Chugai pharmaceutical Co. Ltd.) will be administered subcutaneously at 2- to 6-week interval.
  Dose and interval will be adjusted according to hemoglobin level and its target.
  Arms: High Hb target with cholecalciferol; High Hb target without cholecalciferol
Dietary Supplement: cholecalciferol — 1,000 IU (1 tablet)/day, orally. Tablets are repacked into blister package.
  Other Names: Super vitamin D (Nature Made®)
  Arms: High Hb target with cholecalciferol; Low Hb target with cholecalciferol

SUMMARY:
The purpose of this study is to evaluate the effect of anemia correction and vitamin D supplementation in kidney transplant recipients.

DETAILED DESCRIPTION:
Sample size estimation:

The previous trial (the CAPRIT study) showed that 2.0 g/dL increase of hemoglobin (Hb) reduced 69% of 2-year decline in estimated glomerular filtration rate (eGFR) (Choukroun G, et al. J Am Soc Nephrol, 2012). Given that the annual eGFR decline in our patients with Hb level <10.5 g/dL was 1.66 (SD, 2.47) mL/min per 1.73 m2, the investigators hypothesized that the 2-year eGFR decline in the conservative anemia management group and the aggressive anemia correction group should be 3.32 (SD, 4.94) and 1.03 (SD, 4.94) mL/min per 1.73 m2, respectively. In order to compare the actual efficacy of the intervention with the assumptions above and to evaluate the need for an early termination of the trial, the investigators will perform one interim analysis using a Pocock type α-spending function when a total of 50-60% of the target sample size completed this study or dropped out. Assuming 20% of dropout or lost-to-follow, the planned sample size of 272 patients would yield a power of 90% for group comparison by using t-test with a type I error of 5%.

Regarding cholecalciferol supplementation, 1,000 IU/day would increase serum 25-hydroxyvitamin D level by 11.8 ng/mL in patients with BMI <30, as suggested by the previous trial (Gallagher JC, et al. Ann Intern Med, 2012). The investigators found in our prospective cohort study that the 98.2% of Japanese kidney transplant recipients had BMI <30, and that 10 ng/mL increase in 25-hydroxyvitamin D level was significantly associated with 0.75 mL/min/1.73 m2 less decrease in annual eGFR change independent of potential confounders (in submission). As with the anemia intervention arms above, the investigators will perform one interim analysis using a Pocock type α-spending function when a total of 50-60% of the target sample size completed this study or dropped out in order to compare the actual efficacy of the intervention with the assumptions above and to evaluate the need for an early termination of the trial. Therefore, the investigators expect 1.77 mL/min per 1.73 m2 in eGFR would be preserved by 1,000 IU/day of cholecalciferol supplementation for 2 years. Based on this assumption, this study size will provide a power of 70%.

Estimating kidney function:

In primary analyses, eGFR will be calculated by using the Japanese equation as in sample size calculation (Matsuo S, et al. Am J Kidney Dis, 2009). However, this formula has not yet been validated in kidney transplant recipients. Therefore, the investigators will use the creatinine-based CKD-EPI equation with Japanese coefficient (Stevens LA, et al. Nephrol Dial Transplant, 2010. Horio M, et al. Am J Kidney Dis, 2010) and an available formula if validated in Japanese kidney transplant recipients at the time of analysis.

Statistical analyses:

For group comparison in a primary analysis, the investigators will use t-test or Wilcoxon rank sum test according to the distribution of eGFR change. In the further analyses, to analyze the time course of eGFR with respect to treatment assignment, changes in eGFR over time will be analyzed with a linear mixed model for repeated measures with both fixed and random intercept and slope. The multivariate model will contain time-varying eGFR as dependent variable and treatment group as well as the number of measurements (time) as independent variables. The study hypothesis will be tested by adding appropriate interaction terms between the exposures and time. For secondary endpoints, the investigators will use t-test, Wilcoxon rank sum test, or log-rank test for group comparison, and generalized linear models or Cox proportional hazards models to estimate each effect of the interventions, appropriately. The investigators will also adjust for baseline levels or past history of each outcome. Other potential confounders, such as age, sex, time since transplantation, blood pressure, urinary protein level, and diabetes, will be adjusted in sensitivity analyses.

The interaction will be checked between anemia management and cholecalciferol supplementation as well as between each intervention and baseline levels of urinary protein, eGFR, Hb, 25-hydroxyvitamin D, the use of active vitamin D compounds, and the length of time since transplantation. Additionally, stratified analyses will be conducted according to 0.2 g/g･creatinine of urinary protein and the date of transplantation (November 1999, the release date of mycophenolate mofetil in Japan). However, the study size is not large enough to statistically evaluate these interactions. The results from these analyses should be interpreted with caution and regarded as exploratory and hypothesis generating.

Missing values:

Missing values will not be imputed in primary analyses. In sensitivity analyses, the investigators will use multiple imputation method and last-observation-carried-forward method.

Note:

The interim analysis plan was added to the protocol with an increase in the sample size from 246 to 272, which has been approved by the local ethics committee on August 27, 2018.

ELIGIBILITY:
Inclusion Criteria:

* ≥15 and <60 ml/min per 1.73 m2 of estimated glomerular filtration rate
* Transplanted allograft kidney at least 1 year before
* <10.5 g/dL of Hb without iron deficiency (serum ferritin level ≥50 ng/ml) or on erythropoiesis stimulating agents treatment regardless of iron status
* With written informed consent

Exclusion Criteria:

* On anticancer treatment
* History of ischemic stroke or transient ischemic attack
* Corrected serum calcium ≥10.5 mg/dL
* HIV virus infection
* Anticipated refractory hypertension by using epoetin beta pegol
* In pregnancy and lactation
* Current use of native vitamin D supplement
* Patients ineligible according to the investigator's judgement

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in allograft kidney function | 2 years
  As allograft kidney function, GFR is estimated by the modified MDRD equation for Japanese patients with chronic kidney disease.

SECONDARY OUTCOMES:
Urine markers of kidney injury | 6 months
  1. protein-creatinine ratio
  2. liver type fatty acid binding protein (L-FABP)
  3. neutrophil gelatinase-associated lipocalin (NGAL)
  4. transforming growth factor (TGF)-β.
The dose of methoxy polyethylene glycol epoetin beta required to maintain the target hemoglobin level | 1 year
  For vitamin D supplementation study only.
Blood pressure | 2 years
Cardiac biomarkers | 2 years
  1. brain natriuretic peptide (BNP)
  2. cardiac troponin-T (cTnT).
Left ventricular mass index | 2 years
Biopsy-proven acute cellular rejection | 2 years
Bone-turnover markers | 6 months
  1. intact parathyroid hormone (1-84 PTH)
  2. bone-type alkaline phosphatase
  3. tartrate-resistant acid phosphatase 5b (TRACP-5b)
  For vitamin D supplementation study only.
Bone mineral density of lumber spine and femoral neck. | 2 years
  For vitamin D supplementation study only.
Hypercalcemia | 2 years
  Corrected calcium ≥11 mg/dL
  For vitamin D supplementation study only.
Time to the renal composite endpoint | 2 years
  renal composite endpoint consists of 50% increase in serum creatinine, subsequent transplantation, and reinitiation of dialysis.
Time to admission-required cardiovascular events | 2 years
  Cardiovascular events includes myocardial infarction, angina, congestive heart failure, stroke, and peripheral artery disease.
Time to all-cause death | 2 years
Time to Cancer development or recurrence | 2 years

OTHER OUTCOMES:
C-reactive protein | 1 year
  For vitamin D supplementation study only.
Time to the adverse composite endpoint | 2 years
  The adverse composite endpoint consists of death, admission-required cardiovascular diseases, and the renal composite endpoint.
Time to hospitalization for opportunistic infections | 2 years
  Opportunistic infections includes polyomavirus-associated nephropathy, tuberculosis, Pneumocystis carinii pneumonia, cytomegalovirus infection, herpes zoster, bacterial pneumonia.
  For vitamin D supplementation study only.

CONTACTS AND LOCATIONS:
Overall Officials: Takayuki Hamano, MD, PhD, Study Director — Department of Inter-Organ Communication Research in Kidney Disease, Osaka University Graduate School of Medicine
Locations (1):
- CANDLE Trial Study Group, Suita, Osaka, Japan

REFERENCES:
- [Background] Choukroun G, Kamar N, Dussol B, Etienne I, Cassuto-Viguier E, Toupance O, Glowacki F, Moulin B, Lebranchu Y, Touchard G, Jaureguy M, Pallet N, Le Meur Y, Rostaing L, Martinez F; CAPRIT study Investigators. Correction of postkidney transplant anemia reduces progression of allograft nephropathy. J Am Soc Nephrol. 2012 Feb;23(2):360-8. doi: 10.1681/ASN.2011060546. Epub 2011 Dec 22. PMID 22193388
- [Background] Gallagher JC, Sai A, Templin T 2nd, Smith L. Dose response to vitamin D supplementation in postmenopausal women: a randomized trial. Ann Intern Med. 2012 Mar 20;156(6):425-37. doi: 10.7326/0003-4819-156-6-201203200-00005. PMID 22431675
- [Background] Matsuo S, Imai E, Horio M, Yasuda Y, Tomita K, Nitta K, Yamagata K, Tomino Y, Yokoyama H, Hishida A; Collaborators developing the Japanese equation for estimated GFR. Revised equations for estimated GFR from serum creatinine in Japan. Am J Kidney Dis. 2009 Jun;53(6):982-92. doi: 10.1053/j.ajkd.2008.12.034. Epub 2009 Apr 1. PMID 19339088
- [Background] Stevens LA, Schmid CH, Zhang YL, Coresh J, Manzi J, Landis R, Bakoush O, Contreras G, Genuth S, Klintmalm GB, Poggio E, Rossing P, Rule AD, Weir MR, Kusek J, Greene T, Levey AS. Development and validation of GFR-estimating equations using diabetes, transplant and weight. Nephrol Dial Transplant. 2010 Feb;25(2):449-57. doi: 10.1093/ndt/gfp510. Epub 2009 Sep 30. PMID 19793928
- [Background] Horio M, Imai E, Yasuda Y, Watanabe T, Matsuo S. Modification of the CKD epidemiology collaboration (CKD-EPI) equation for Japanese: accuracy and use for population estimates. Am J Kidney Dis. 2010 Jul;56(1):32-8. doi: 10.1053/j.ajkd.2010.02.344. Epub 2010 Apr 22. PMID 20416999